CLINICAL TRIAL: NCT05458531
Title: Exploring Patient and Healthcare Professional Views and Experiences of the Current and Recommended Monitoring Strategies for Inflammatory Conditions Treated With Commonly Used Immune Suppressing Drugs
Brief Title: Monitoring of Inflammatory Conditions
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 21042
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Inflammatory Disease; Crohn Disease; Ulcerative Colitis; Rheumatoid Arthritis; System; Lupus Erythematosus; Psoriatic Arthritis; Reactive Arthritis; Inflammatory Arthritis; Psoriasis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Arthritis, Psoriatic; Arthritis, Reactive; Arthritis; Psoriasis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with an inflammatory disease taking immune-suppressing medication: Aged 18 years and over, able to give consent, diagnosed with one of the above inflammatory conditions and currently treated with one of the following immune-suppressing treatments for six months or longer: methotrexate, azathioprine, 5-acetyl salicylates, sulfasalazine, mycophenolate mofetil, leflunomide or biologics.
  Interventions: Other: Questionnaire; Other: Semi-structured interview
- Healthcare professionals: Consultants, general practitioners (GPs), nurse specialists, practice nurses and pharmacists with experience of prescribing and monitoring long-term immune-suppressing treatments for the above inflammatory diseases
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Questionnaire — A single questionnaire
  Groups: Patients with an inflammatory disease taking immune-suppressing medication
Other: Semi-structured interview — A single semi-structured qualitative interview conducted face-to-face or by telephone or video-conference call.

SUMMARY:
People with inflammatory diseases treated with immune-suppressing medication are recommended to have regular blood-tests to monitor for potential side-effects of this treatment on their blood count, liver and kidneys. However, it is not clear that monitoring is needed as frequently as currently recommended in the long-term, with side-effects being rare after one year of treatment. A study is currently underway to determine the optimal blood-test monitoring strategy which is cost-effective but still safe. Any changes in the monitoring strategy must be acceptable to patients and the healthcare professionals (HCP) that treat them.

This study aims to measure how often patients' with common inflammatory conditions on long-term immune suppressing medication attend their monitoring blood tests as currently recommended, and uncover patients' and HCP views and experiences of the current blood-test monitoring strategy, and the acceptability of potential changes to this in the future.

Firstly, patients with an inflammatory condition on long-term immune suppressing treatment will be invited to complete a questionnaire which will ask about their demographic information, medical condition(s), immune-suppressing treatment, adherence to the monitoring blood tests and willingness to take part in an interview. Then, both patients and HCPs who care for such patients will be invited to take part in a single, semi-structured interview. Interviews will be face-to-face, by telephone or video-call, last up to one hour and digitally audio-recorded. Patient interviews will explore their perceptions of risk, benefits and experiences of current testing, and views on the new testing frequencies emerging from the study prior. HCP interviews will explore their perceptions of current testing including, the practicalities, usefulness, risks and benefits of the blood tests, and views on the new testing frequencies emerging from the study prior.

The findings will shape the recommendations for a new monitoring strategy, ensuring it is acceptable to patients and HCPs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over
* Ability to give informed consent
* Diagnosis with one of the following inflammatory diseases: rheumatoid arthritis, inflammatory arthritis, inflammatory bowel disease, psoriasis +/- arthritis, ankylosing spondylitis, systemic lupus erythematosus, or reactive arthritis, and
* Currently treated with one of the following immune suppressing treatments for six months or longer: methotrexate, azathioprine, 5-acetyl salicylates, sulfasalazine, mycophenolate mofetil, leflunomide or biologics (anti-TNF-α agents e.g. etanercept, adalimumab, infliximab, golimumab, or certolizumab or their biosimilar).

Exclusion Criteria:

* Chronic kidney disease: stage 4 or stage 5
* Chronic liver disease: Autoimmune hepatitis, hepatitis B or C, cirrhosis.
* Pre-existing haematological abnormalities: Myelodysplasia, primary haematological diseases with neutropenia or thrombocytopenia.
* Dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Secondary care clinic and general population
Sampling Method: Non-Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
To explore patient and HCP views and experiences of the current monitoring strategies. | 1 day
  This will be determined through interview
To measure patient adherence with current monitoring recommendations. | 1 day
  This will determined through patient questionnaire
To explore the acceptability of the new recommended monitoring strategy emerging from a prior modelling exercise, to patients and HCPs. | 1 day
  This will be determined through interview

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Abhishek, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No